CLINICAL TRIAL: NCT02697123
Title: Prospective Assessment of the Deep Vein Thrombosis (DVT) in Hospitalized Obstetrics Patients
Status: Terminated | Type: Observational
Why Stopped: PI is no longer at the institution
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael A Belfort, Professor and Chair, Baylor College of Medicine
Other Study IDs: H-36192
Record Dates: First submitted 2016-02-25; First posted 2016-03-03 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Venous Thrombosis; Pregnancy
Keywords: Venous Thrombosis; Pregnancy; postpartum; antepartum
MeSH Terms: conditions — Venous Thrombosis | interventions — Postpartum Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- antepartum and postpartum: This prospective, observational cohort study was designed to assess the incidence of VTE in patients hospitalized for Cesarean Section, Vaginal delivery or any antepartum indication.
  Interventions: Other: antepartum and postpartum

INTERVENTIONS:
Other: antepartum and postpartum — This is a prospective observational cohort study.

SUMMARY:
The purpose of the study is to prospectively assess the prevalence of venous thrombosis in women hospitalized for Cesarean Section, vaginal delivery or extended antepartum hospitalization by using Compression ultrasound of the entire proximal venous system of the lower limb veins.

DETAILED DESCRIPTION:
After initial admission of the patients for Cesarean Section, Vaginal Delivery or any other antepartum hospitalization, patients undergo extensive counseling regarding various aspects of the Duplex Ultrasonography procedure and the purpose of the study for screening of the venous thrombosis in asymptomatic patients. Patients electing to proceed will have written informed consent obtained and their baseline demographic and medical characteristics recorded. 48-72 hours after Cesarean Section, 24-48 hours after vaginal delivery and 48 to 72 hours after antepartum hospitalization, participants also undergo a bilateral lower extremity Venous Ultrasonographic examination which is the standard diagnostic procedure for detecting the VTE of the lower limbs. The latter group will be re-scanned 14-21 days and, when feasible, 45 days after admission.

The compression ultrasound study will be performed by post-doctoral research fellows, who will be formally trained for lower extremity ultrasound, under direct supervision. Diagnostic Criteria and Interpretation · The gray scale compression sonographic findings of acute DVT are based on direct visualization of the thrombus and lack of venous compressibility. Altered luminal echogenicity and alterations in flow characteristics are secondary signs. · Visualization of thrombus is variable, depending on the extent, age, and echogenicity (ranging from anechoic to complex) of the clot. · in case of thrombosis, Each Doppler image should demonstrate spontaneous and phasic flow. · Loss of phasic variation suggests proximal obstruction (intrinsic or extrinsic). · Prominent pulsations can be due to right sided heart failure and may be a manifestation of tricuspid valve regurgitation. Normal - Vein is totally compressible. Duplex Doppler reveals spontaneous phasic waveform Acute DVT - Vein is non compressible, but deformable and smooth. Vein is generally distended, with or without luminal echoes. The thrombus can be free floating. Spectral Doppler may be normal, continuous, or not present

If no DVT is seen on ultrasonography, then participants will be followed up clinically throughout the remainder of their hospitalization without further intervention. Participants with a DVT in the deep venous circulation will be referred to radiology for confirmation and if positive for DVT the patient will be offered treatment per current clinical guidelines for symptomatic DVT. This was the approach taken in most similar studies involving detection of DVT in asymptomatic non-pregnant women.

If a VTE is seen in the superficial veins of the lower extremity, another lower extremity venous Ultrasonographic evaluation will be scheduled 48 hours later. If a persistent superficial VTE is seen, the patient will be referred for evaluation and therapy per current clinical guidelines.

Ultrasound procedure data and all the information related to the findings of this study like the reports, ultrasound pictures or demographic informations will be stored in the subject's medical records which will be created specifically for this study.

All the imaging will be reviewed blindly by one sonographer and one radiologist for image quality. If the image is not qualified and patient is still at hospital will redo the Doppler ultrasound. if the patient is discharged will exclude that patient from the study.

We will also collect demographic data and other clinical information of the patient such as maternal age, prenatal records, ultrasounds reports at different gestational age, consultations, maternal past medical history, maternal past obstetrical history, medications receive during pregnancy, gestational age at the time of procedure, first manifestation of the DVT, treatments, process of these conditions, outcome, gestational age at birth, fetal anomalies, early neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized for Cesarean Section,
* All patients hospitalized for vaginal delivery
* any other antepartum indication of hospitalization.

Exclusion Criteria:

* Psychiatric illness
* social situations that could limit compliance with study activities
* all patients who lack capacity to consent.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients presenting to TCH/Women's Pavilion and Ben Taub Hospital for Cesarean Section, vaginal delivery or any antepartum hospitalization will considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
incidence of Venous Thrombosis in patients hospitalized for Cesarean Section, Vaginal delivery or any antepartum indication | 48 hours (plus or minus 24 hours) after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Clark, M.D., Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided